CLINICAL TRIAL: NCT00579007
Title: Decision-making Regarding Prophylactic Mastectomy and Oophorectomy in Women Seeking Genetic Counseling and Testing for BRCA1/2 Mutations
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 03-001
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Prophylactic Mastectomy; Prophylactic Oophorectomy
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women with a strong family history of breast cancer.
  Interventions: Behavioral: telephone interviews

INTERVENTIONS:
Behavioral: telephone interviews — Telephone interviews take place before the first counseling appointment (baseline), and 1 week, 6 months and 12 months post-notification of the individual's genetic test results. In the event that a participant chooses not to undergo genetic testing, follow-up interviews will take place 1 month, 6 months and 12 months after the initial counseling visit.

SUMMARY:
The purpose of this study is to learn more about women's decision to undergo prophylactic surgery. This is removal of healthy organs in order to reduce risk of cancer. This study will help us to understand what makes women decide whether or not to have this kind of surgery.

DETAILED DESCRIPTION:
For women with a strong family history of breast/ovarian cancer, few options exist for primary prevention of these cancers other than prophylactic surgery, or surgical removal of noncancerous organs in order to prevent occurrence of the disease. The primary aim of the study is to describe the stages of intention to undergo prophylactic mastectomy and/or oophorectomy among women seeking genetic testing for inherited BRCA1 and BRCA2 mutations, and to identify factors that influence stages of intention regarding prophylactic surgery. To achieve these aims, 626 women undergoing genetic counseling and testing for inherited breast ovarian cancer risk will be assessed before their first genetic counseling session and three times (1 week, 6 months and 12 months) in the year following notification of their genetic test results.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* age 25 and above
* a personal or family history of breast and/or ovarian cancer showing clinical features associated with increased risk of carrying a BRCA1/2 mutation (e.g., breast and ovarian cancer on the same side of the family, early age of onset, multiple primaries in the same individual) or having a first-degree relative with a known BRCA1 or BRCA2 mutation.

Exclusion Criteria:

* Male gender
* age less than 25 years
* unable to provide meaningful informed consent due to physical, cognitive or psychiatric disability
* non-English speaking

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing genetic counseling and testing for inherited breast or ovarian ccancer risk will be assessed before their first genetic counseling session
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2003-03-11 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Primary outcome of the study is stage of intention to undergo prophylactic surgery. Outcome variable consists of 6 rank-ordered, qualitatively distinct stages (see Measures) ranging from Precontemplation (no intention) to Action (intention carried out). | 1 year

SECONDARY OUTCOMES:
To determine the relative contributions of sociodemographic, medical, and psychosocial factors to stage of intention regarding prophylactic mastectomy and/or oophorectomy. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Lichtenthal, Ph.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org